CLINICAL TRIAL: NCT01144520
Title: Leukocyte Dysfunction in Diabetic Patients.
Status: Terminated | Type: Observational
Why Stopped: researchers moved to new institution and did not transfer project
Sponsor: Sashwati Roy (Other)
Responsible Party: Sponsor-Investigator, Sashwati Roy, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2009H0270
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normoglycemic: Healthy subjects that do not have diabetes
- Type II Diabetes (HbA1c <7 or 7%): Subject that have Type II Diabetes with good glucose control with glycated hemoglobin (HbA1c <7 or 7%)
- Type II Diabetes (HbA1c between 7.1-9): Subjects with Type II Diabetes with moderate glucose control (HbA1c between 7.1-9)
- Type II Diabetes (HbA1c >9%): Subjects with Type II Diabetes with poor glucose control (HbA1c >9%)

SUMMARY:
The purpose of this study is to study impairment of white blood cell function in patients with type II diabetes.

DETAILED DESCRIPTION:
Leucocytes from poorly controlled diabetes exhibit aberrant chemotaxis, increased susceptibility to bacterial infection, leukotriene production, lysosomal enzyme release, proinflammatory cytokine expression and production of reactive oxygen species. Aberrant glucose concentration in diabetics affects functions of peripheral blood system as well as the immune system leading to impaired host defense. Impaired wound healing is a serious complication associated with diabetes. We hypothesized that impairment in leukocyte function results in dysfunctional inflammatory response in diabetic wounds. The proposed studies focus on characterizing mechanisms that will improve our understanding of the dysfunctional inflammatory response resulting in non-healing chronic wounds in diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 40-60 yrs old clinically diagnosed with Type II Diabetes
* Adults ages 40-60 yrs old without Diabetes

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant Females
* Therapeutically Immuno-compromised

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the population who visit the Ohio State University (OSU) Hospitals and Comprehensive Wound Center (CWC), OSU Wexner Medical Center diabetic clinics and Bariatric clinic.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Ex vivo leukocyte function by measuring ROS production | immediately after blood draw
  After blood draw monocytes are separated from whole blood and production of oxidants by these cells

SECONDARY OUTCOMES:
Ex vivo NADPH oxidase gene and protein expression | After blood draw
  Gene and protein expressions are measured using Western blot and real time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Sashwati, MS, PhD, Principal Investigator — Ohio State University Dept of Surgery
Locations (1):
- Ohio State University Comprehensive Wound Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Shurtz-Swirski R, Sela S, Herskovits AT, Shasha SM, Shapiro G, Nasser L, Kristal B. Involvement of peripheral polymorphonuclear leukocytes in oxidative stress and inflammation in type 2 diabetic patients. Diabetes Care. 2001 Jan;24(1):104-10. doi: 10.2337/diacare.24.1.104. PMID 11194213
- [Result] Lin X, Candlish JK, Thai AC. Superoxide production by neutrophils from diabetics and normal subjects in response to glucose and galactose. Exp Mol Pathol. 1993 Jun;58(3):229-36. doi: 10.1006/exmp.1993.1020. PMID 8390941
- [Result] Molenaar DM, Palumbo PJ, Wilson WR, Ritts RE Jr. Leukocyte chemotaxis in diabetic patients and their nondiabetic first-degree relatives. Diabetes. 1976;25(2 SUPPL):880-3. PMID 971792
- [Result] Hill HR, Sauls HS, Dettloff JL, Quie PG. Impaired leukotactic responsiveness in patients with juvenile diabetes mellitus. Clin Immunol Immunopathol. 1974 Apr;2(3):395-403. doi: 10.1016/0090-1229(74)90057-9. No abstract available. PMID 4826528
- See also: OSU Center for Regenerative Medicine and Cell Based Therapies — http://medicine.osu.edu/regenerativemedicine/Pages/index.aspx
- See also: OSU Comprehensive Wound Center — http://medicalcenter.osu.edu/patientcare/healthcare_services/wound_care/Pages/index.aspx